CLINICAL TRIAL: NCT01561521
Title: An Evaluation of the Onset and Duration of Action of AKF-1 Ophthalmic Solution in Treating Acute Allergic Conjunctivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Akorn, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11-100-0008
Record Dates: First submitted 2012-03-21; First posted 2012-03-23 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2012-05

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- AKF-1 0.025% (Experimental)
  Interventions: Drug: AKF-1
- AKF-1 0.035% (Experimental)
  Interventions: Drug: AKF-1
- AKF-1 0% (Placebo Comparator)
  Interventions: Drug: AKF-1

INTERVENTIONS:
Drug: AKF-1 — 1 drop AKF-1 0.025% in each eye at 2 separate times during a 14 day period
  Arms: AKF-1 0.025%
Drug: AKF-1 — 1 drop AKF-1 0.035% in each eye at 2 separate times during a 14 day period
  Arms: AKF-1 0.035%
Drug: AKF-1 — 1 drop 0% in each eye at 2 separate times during a 14 day period
  Arms: AKF-1 0%

SUMMARY:
The purpose of this study is to evaluate the onset and duration of action of two concentrations of AKF-1 Ophthalmic Solution compared to vehicle in the conjunctival allergen challenge (CAC) model of acute allergic conjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* positive bilateral conjunctival allergen challenge (CAC) reaction

Exclusion Criteria:

* known contraindications or sensitivities to the study medication or its components
* any ocular condition that, in the opinion of the investigator, could affect the subjects safety or trial parameters
* use of disallowed medication during the period indicated prior to the enrollment or during the study

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2012-03; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Ocular Itching at defined time points up to 2 weeks | Baseline to day 14
Ocular Redness at defined time points up to 2 weeks | Baseline to day 14

CONTACTS AND LOCATIONS:
Locations (1):
- Andover Eye Associates, Andover, Massachusetts, United States